CLINICAL TRIAL: NCT00510406
Title: A Randomized, Double-blind, Parallel Group, Placebo Controlled, Multi Center Dose Ranging Study of Solifenacin Succinate in Combination With Tamsulosin Hydrochloride Compared With Solifenacin Succinate Monotherapy and Tamsulosin Hydrochloride Monotherapy in Males With Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH)
Brief Title: A Study With Combination Treatment (Tamsulosin Hydrochloride and Solifenacin Succinate) in Male Patients With LUTS/BPH
Acronym: SATURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-CL-052; EudraCT number: 2006-002072-18
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Lower Urinary Tract Symptoms; Prostatic Hyperplasia
Keywords: Lower Urinary Tract Symptoms; Treatment; Solifenacin succinate; Tamsulosin hydrochloride; Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Active Comparator)
  Interventions: Drug: solifenacin succinate
- C (Active Comparator)
  Interventions: Drug: solifenacin succinate
- D (Active Comparator)
  Interventions: Drug: solifenacin succinate
- E (Active Comparator)
  Interventions: Drug: tamsulosin hydrochloride
- F (Active Comparator)
  Interventions: Drug: tamsulosin hydrochloride; Drug: solifenacin succinate
- G (Active Comparator)
  Interventions: Drug: tamsulosin hydrochloride; Drug: solifenacin succinate
- H (Active Comparator)
  Interventions: Drug: tamsulosin hydrochloride; Drug: solifenacin succinate

INTERVENTIONS:
Drug: tamsulosin hydrochloride — Alphablocker
  Arms: E; F; G; H
Drug: solifenacin succinate — antimuscarinic
  Arms: B; C; D; F; G; H
Drug: Placebo — Placebo
  Arms: A

SUMMARY:
The study will examine the efficacy,safety and tolerability of combination therapy of tamsulosin and solifenacin compared to placebo and monotherapy of tamsulosin and solifenacin in the treatment of males with LUTS associated with BPH.

DETAILED DESCRIPTION:
Placebo Solifenacin succinate Tamsulosin hydrochloride Tamsulosin hydrochloride + solifenacin succinate

The primary comparison will be the combination treatment with tamsulosin hydrochloride monotherapy.

Other comparisons will be:

Placebo and combination treatment. Solifenacin monotherapy and combination treatment

ELIGIBILITY:
Inclusion Criteria:

* male patients with LUTS associated with BPH diagnosed > 3 months
* IPSS score > 13
* voiding and storage symptoms
* maximum flow rate of > 4 mL/s and < 15 mL/s

Exclusion Criteria:

* post void residual volume > 200 mL
* symptomatic urinary tract infection

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Assess whether the combination of solifenacin succinate and tamsulosin hydrochloride provides improved efficacy compared to tamsulosin hydrochloride alone in males with LUTS associated with BPH | 12 weeks

SECONDARY OUTCOMES:
Assess efficacy, safety, tolerability and PK of the combination of solifenacin succinate and tamsulosin hydrochloride | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (98):
- Austria (3):
  - Linz, North-West
  - Graz, Styria
  - Vienna, Vienna
- Czechia (4):
  - Ostrava
  - Pilsen
  - Prague
  - Ústí nad Labem
- Denmark (4):
  - Aalborg
  - Frederiksberg
  - Roskilde
  - Skejby
- Finland (5):
  - Helsinki
  - Kuopio
  - Lahti
  - Oulu
  - Tampere
- France (9):
  - Colmar
  - Cote de Nacre
  - Créteil
  - Marseille
  - Montluçon
  - Mulhouse
  - Nîmes
  - Paris
  - Ploemeur
- Germany (18):
  - Bad Segeberg
  - Bamberg
  - Bautzen
  - Dresden
  - Eisleben Lutherstadt
  - Ganderkessee
  - Hagenow
  - Halle
  - Hamburg
  - Henningsdorf
  - Hettstedt
  - Koblenz
  - Leipzig
  - München
  - Münster
  - Neustadt in Sachsen
  - Trier
  - Uetersen
- Hungary (8):
  - Budapest
  - Eger
  - Miskolc
  - Nyiregyháza
  - Sopron
  - Szeged
  - Szekszárd
  - Tatabánya
- Netherlands (9):
  - Nijmegen, Gelderland
  - Maastricht, Limburg
  - S'Hertogenbosch, North Brabant
  - Tilburg, North Brabant
  - Amsterdam, North Holland
  - Apeldoorn, Overijssel
  - Deventer, Overijssel
  - Sneek, Provincie Friesland
  - Utrecht, Utrecht
- Norway (3):
  - Fredrikstad
  - Oslo
  - Tønsberg
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Katowice
  - Krakow
  - Lódz
  - Lublin
  - Puławy
  - Szczecin
  - Warsaw
- Portugal (7):
  - Amadora-Sintra
  - Carmo
  - Coimbra (Covões)
  - Orta EPE
  - Pulido Valente
  - Santa Luzia
  - Tomar
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (3):
  - Nitra
  - Trenčín
  - Žilina
- Spain (5):
  - A Coruña
  - Barcelona
  - Madrid
  - Pontevedra
  - Seville
- Sweden (5):
  - Kungälv
  - Stockholm
  - Sundsvall
  - Uddevalla
  - Uppsala
- United Kingdom (4):
  - Reading, Berkshire
  - Chorley, Lancashire
  - Cardiff, Wales
  - Swansea, Wales

REFERENCES:
- [Derived] Van Kerrebroeck P, Haab F, Angulo JC, Vik V, Katona F, Garcia-Hernandez A, Klaver M, Traudtner K, Oelke M. Efficacy and safety of solifenacin plus tamsulosin OCAS in men with voiding and storage lower urinary tract symptoms: results from a phase 2, dose-finding study (SATURN). Eur Urol. 2013 Sep;64(3):398-407. doi: 10.1016/j.eururo.2013.03.031. Epub 2013 Mar 19. PMID 23537687